CLINICAL TRIAL: NCT05598320
Title: A Phase 2b, Multicenter, Double-Blind, Randomized, Placebo-controlled Trial Evaluating Efficacy and Safety of Subcutaneous Doses of TransCon CNP Administered Once Weekly for 52 Weeks in Children With Achondroplasia Followed by an Open Label Extension Period
Brief Title: A Clinical Trial to Evaluate Efficacy and Safety of TransCon CNP Compared With Placebo in Children With Achondroplasia
Acronym: ApproaCH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ascendis Pharma Growth Disorders A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASND0036
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TransCon CNP (Experimental): Once weekly double-blinded treatment with SC injection of 100 µg/kg of TransCon CNP for 52 weeks
  Interventions: Drug: TransCon CNP
- Placebo for TransCon CNP (Placebo Comparator): Once weekly double-blinded treatment with SC injection of 100 µg/kg of Placebo for TransCon CNP for 52 weeks
  Interventions: Drug: Placebo for TransCon CNP
- Open-Label Extension Period: TransCon CNP (Experimental): Participants who completed the 52-week blinded treatment period continued into the open-label extension period and received treatment with TransCon CNP 100 µg/kg delivered once weekly by subcutaneous injection.
  Interventions: Drug: TransCon CNP

INTERVENTIONS:
Drug: TransCon CNP — Once-weekly subcutaneous injection of 100 µg/kg TransCon CNP
  Arms: Open-Label Extension Period: TransCon CNP; TransCon CNP
Drug: Placebo for TransCon CNP — Once-weekly subcutaneous injection of 100 µg/kg placebo for TransCon CNP
  Arms: Placebo for TransCon CNP

SUMMARY:
The purpose of this clinical trial is to evaluate efficacy and safety of once weekly SC doses of 100 µg CNP/kg compared to placebo on Annualized Growth Velocity after a 52-week randomized treatment period in children aged 2 to 11 years with genetically confirmed Achondroplasia. The double-blind, placebo-controlled treatment period is followed by an Open Label Extension (OLE) period of a 52-week duration.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed informed consent of the parent(s) or legal guardian(s) of the participant, and as required by the institutional review board/human research ethics committee/independent ethics committee (IRB/HREC/IEC).
* Male or female, between 2 and 11 years of age (inclusive) at the time of Screening.
* Clinical diagnosis of ACH with documented genetic confirmation available.
* Able to stand without assistance.
* Parent(s)/legal guardian(s) willing and able to administer weekly SC injections of IMP and to follow the protocol.
* At least six months of growth and disease history from ACHieve (TCC-NHS-01) trial or comparable growth and disease history available from medical records (pending confirmation by Medical Monitor).
* Considered eligible based on the medical history, physical examination, and the results of vital signs, ECG and clinical laboratory tests performed during the Screening period

Exclusion Criteria:

* Participation (i.e., signed informed consent) in any interventional clinical trial before within 3 months prior to screening.
* Closed epiphysis.
* Known or suspected hypersensitivity to the IMP or related products (trehalose, tris[hydroxymethyl]aminomethane, succinate, and mPEG).
* Have a growth disorder or medical condition other than ACH that results in short stature or abnormal growth such as severe ACH with developmental delay and acanthosis nigricans (SADDAN), hypochondroplasia, growth hormone deficiency, Turner syndrome, pseudoachondroplasia, inflammatory bowel disease, celiac disease, hypothyroidism, hyperthyroidism, pre-diabetes, or diabetes mellitus.
* Have received any dose of prescription medications and IMP or surgical intervention intended to affect stature, growth, or body proportionality at any time.
* Requires, or anticipated to require, chronic (> 4 weeks) or repeated treatment (more than twice/year and >3 weeks/year) with systemic corticosteroids during participation in the trial. Chronic use of high-dose inhaled corticosteroids is not allowed.
* Known history of presence of injury or disease of the growth plate(s), other than ACH, that affects growth potential of long bones.
* Known history of any bone-related surgery affecting growth potential of long bones, such as:

  * Orthopedic reconstructive surgery for bone lengthening (e.g., procedures for leg bowing such as 8-plate are not exclusionary).
  * Cervicomedullary decompression surgery without anticipated need for repeat decompression during the time of the trial are allowed with minimum of 6 months of bone healing.
  * Ventriculoperitoneal (VP) shunt and laminectomy with full recovery are allowed with minimum of 6 months of bone healing.
  * Bone fracture within 6 months prior to screening (within 2 months for fracture of digits and buckle fractures).
* Clinically significant findings at Screening, such as:

  * Expected to require surgical intervention during participation in the trial. Common surgeries, such as insertion of grommets, adenoidectomy, tonsillectomy, or myringotomy tube placement, are permitted.
  * Severe untreated sleep apnea or newly initiated sleep apnea treatment (e.g., Continuous Positive Airway Pressure [CPAP] in the previous 2 months prior to Screening).
  * Musculoskeletal disease, such as Salter-Harris fractures or clinical and/or radiographic evidence of severe hip pathology, or
  * Otherwise, are considered by the Investigator and Medical Monitor to make a participant unfit to receive trial treatment or undergo trial related procedures.
* Have evidence at Screening that are consistent with severe cervicomedullary junction compression based on clinical and/or radiologic findings that indicate immediate surgical intervention is required.
* Have a clinically significant finding or arrhythmia as determined by the investigator in consultation with the medical monitor that indicates abnormal cardiac function or conduction that includes, but is not exclusive to:

  * Repaired or unrepaired coarctation.
  * Moderate or greater complexity congenital heart disease including tetralogy of Fallot, Atrioventricular septal defects, truncus arteriosus, total anomalous pulmonary venous return, double outlet right ventricle, or single ventricle heart disease.
* QTcF ≥ 450 msec at the Screening Visit.
* Known history or presence of condition that impacts hemodynamic stability (such as autonomic dysfunction and orthostatic intolerance).
* Known history or presence of the following:

  * Chronic anemia (iron deficiency anemia that is resolved or adequately treated in the Investigator's opinion is allowed).
  * Chronic renal insufficiency (GFR <60 mL/min/1.73 m2 for >3 months).
  * Chronic or recurrent illness that can affect hydration or volume status, including conditions associated with decreased nutritional intake or increased volume loss.
* Known history or presence of malignant disease.
* Participant with serum 25-hydroxy-vitamin D (25OHD) levels of <30 nmol/L (<12 ng/mL) at Screening Visit will be excluded. Participants with 25OHD levels between 30-50 nmol/L (12-20 ng/mL) can be randomized provided treatment with Vitamin D supplementation is initiated.
* Any disease or condition that, in the opinion of the Investigator, may make the participant unlikely to fully complete the trial, may confound interpretation of trial results, or may present undue risk from receiving trial treatment. This could include family situations, complications or manifestations, or medications that might impact safety or be considered confounding.
* Sexually active male and female participants and female partners of male participants of childbearing potential not using a highly effective form of contraceptive for the entire trial period and for 90 days after last dose of trial treatment.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Annualized Growth Velocity | 52 weeks
  cm per year

SECONDARY OUTCOMES:
Height Z-score | 52 weeks
  Number of standard deviations

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Ascendis Pharma A/S
Locations (10):
- United States (4):
  - Ascendis Pharma Investigational Site, Saint Paul, Minnesota
  - Ascendis Pharma Investigational Site, Columbia, Missouri
  - Ascendis Pharma Investigational Site, Houston, Texas
  - Ascendis Pharma Investigational Site, Madison, Wisconsin
- Ascendis Pharma Investigational Site, Parkville, Australia
- Ascendis Pharma Investigational Site, Montreal, Canada
- Ascendis Pharma Investigational Site, Copenhagen, Denmark
- Ascendis Pharma Investigational Site, Dublin, Ireland
- Ascendis Pharma Investigational Site, Auckland, New Zealand
- Ascendis Pharma Investigational Site, Vitoria-Gasteiz, Spain

IPD SHARING:
Plan to Share IPD: No
Not planned

REFERENCES:
- [Derived] Savarirayan R, McDonnell C, Bacino CA, Hoernschemeyer DG, Legare JM, Abuzzahab MJ, Hofman PL, Campeau PM, de Bergua Domingo JM, Ward LM, Smit K, Smith A, Mao M, Ominsky MS, Freiberg LC, Shu AD, Hove HB. Once-Weekly Navepegritide in Children With Achondroplasia: The APPROACH Randomized Clinical Trial. JAMA Pediatr. 2026 Jan 1;180(1):18-25. doi: 10.1001/jamapediatrics.2025.4771. PMID 41247754